CLINICAL TRIAL: NCT03149965
Title: Maternal Body Mass Index and Anovaginal Distance in Active Phase of Labor at Term Pregnancy
Brief Title: Maternal Body Mass Index and Anovaginal Distance
Acronym: AVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marie Blomberg, Associated professor, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 930209ec
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Pregnancy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body mass index 18.5-24.9 (Active Comparator): The anovaginal distance was measured with transperineal ultrasound. The standardized method consisted of placing the vaginal probe at a right angle to the posterior vaginal distal wall, and in a transversal scanning plane. The internal anal sphincter was detected as a low-echogenic ring when the probe was moved cranially from the distal anal canal to the mid anal canal. The anovaginal distance was defined as the distance between the anal mucosa and the vaginal wall at the middle level of the anal.
  Interventions: Other: transperineal ultrasound
- body mass index ≥30 (Experimental): The anovaginal distance was measured with transperineal ultrasound. The standardized method consisted of placing the vaginal probe at a right angle to the posterior vaginal distal wall, and in a transversal scanning plane. The internal anal sphincter was detected as a low-echogenic ring when the probe was moved cranially from the distal anal canal to the mid anal canal. The anovaginal distance was defined as the distance between the anal mucosa and the vaginal wall at the middle level of the anal.
  Interventions: Other: transperineal ultrasound

INTERVENTIONS:
Other: transperineal ultrasound — transperineal ultrasound was used by placing a vaginal ultrasound probe towards the vaginal distal wall pointing to the anus, measuring the anovaginal distance.

SUMMARY:
The hypothesis was that the anovaginal distance (AVD), defined as the distance between the anal mucosa and the vaginal wall at the middle level of the anal canal, is higher in obese women compared with normal weight women. Measuring the AVD with transperineal ultrasound has been shown to have a high interobserver agreement.

This study aimed to establish if there was a difference in AVD measured by transperineal ultrasound between obese and normal weight women in active phase of labor at term pregnancy. The second aim was to present normal values for the AVD in active phase of labor at term pregnancy.

DETAILED DESCRIPTION:
This is a prospective cohort study including primiparous women in active phase of labor at term pregnancy on admission at the delivery ward at Linkoping University hospital. The study period was between October 2014 and March 2016. Term pregnancy was defined as ≥ 37 - ≤ 42 gestational weeks. The women had to be in active labor according to the Swedish definition; two out of three of the following criteria must be present: painful contractions (two to three contractions in every ten minutes), cervix shortened and dilated > one centimeter (cm) and/or rupture of membranes. The maximum cervix dilatation allowed for inclusion was seven cm. Further the participant had to be proficient in the Swedish language and aged ≥18 years. All participants were given written and verbal information of the study. The verbal consent to participate was documented in the women´s medical record.

A total number of 207 women were included in the study. There was no information available about whether the women declined participation or if they were not invited to participate. 333 women were excluded due to prematurity, cervix dilatation > seven cm when the women were signed in at the delivery ward, younger than 18 years or not speaking satisfactory Swedish language. After woman's informed consent, the AVD was measured with transperineal ultrasound. The standardized method consisted of placing the vaginal probe at a right angle to the posterior vaginal distal wall, and in a transversal scanning plane. All examinations were done with the patient in the lithotomy position. The internal anal sphincter was detected as a low-echogenic ring when the probe was moved cranially from the distal anal canal to the mid anal canal. The AVD in this study was measured and defined as the distance between the anal mucosa and the vaginal wall at the middle level of the anal canal. The measured AVD, in millimeters (mm), was documented in the women´s medical record under a specific keyword named "anovaginal distance".

The examiners had different proficiency in vaginal ultrasound. As a minimum training to be allowed to include women in the study, the midwives and doctors were trained individually in a defined education program. The education program was based on co-measuring the AVD with one of two experienced experts of AVD-measurement ( ref metodartikeln) . All examiners had to perform co-measurements in at least five women in term pregnancy. Each woman was, after informed consent, measured three times by both the expert and the examiner at education. These women were not included in the present study. The measured AVD values were not shared by the expert and the examiner. The AVD values were compared afterwards, outside the delivery room. In order to be given permission to independently measure the AVD, the examiners had to perform similar values (+/- five mm) as the expert, in five women. Proficiency was achieved among all examiners.

Information on measured AVD, maternal age, smoking status in early pregnancy, ethnicity, measured maternal weight and maternal height in early pregnancy was extracted from the digitalized medical records for every participant and manually registered in an anonymous research database. Gestational weight gain was defined as the difference between the registered weight in kilograms (kg) at the first antenatal visit to the antenatal care center, and the registered weight in term pregnancy at the delivery ward. If there was no registered weight at the delivery ward, the last registered weight at the antenatal care center (between gestational week 37-42) was used to calculate gestational weight gain.

The study population was then divided into three Body Mass Index (BMI) classes based on measured maternal weight and height in early pregnancy (gestational week 10-12); normal weight (BMI <25) , overweight (BMI 25-29.9) and obese (BMI ≥30) . Maternal obesity (BMI ≥30) was also subdivided into obesity class I (BMI 30-34.9) obesity class II (BMI 35-39.9) and obesity class III (BMI ≥40) as suggested by WHO.

The number of women included was based on a power calculation where the relevant difference in AVD between the BMI groups was set to be 10 mm and significance level were equals five percent. A stipulation that a difference of five mm in the AVD could be of clinical relevance was performed. The sample size in each BMI group was calculated to be at least 30 to reach a power of 80% to detect five mm difference in the AVD.

Statistical analyses were performed in order to compare background characteristics between different BMI groups using One-way Anova for continuous variables and X2-test for categorical variables. Post hoc tests were adjusted by the method of Tukey. A two-way Anova was used in order to analyze BMI groups and measurer simultaneously. A p-value of <0.05 was considered significant. Statistical analyses were performed using the Statistical Package for the Social Sciences (IBM SPSS Statistics, Chicago, IL, USA; version 22)

ELIGIBILITY:
Inclusion Criteria:

* Active labor according to the Swedish definition; two out of three of the following criteria must be present: painful contractions (two to three contractions in every ten minutes), cervix shortened and dilated > one centimeter (cm) and/or rupture of membranes.
* The maximum cervix dilatation was of seven centimeters.
* The participant had to be aged ≥18 years
* The participant had to be proficient in the Swedish language

Exclusion Criteria:

* Not in active labor,
* Cervix dilatation of more than seven centimeters,
* Age <19
* Not speaking Swedish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 207 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
anovaginal distance | five minutes
  millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Marie Blomberg, Assoc prof, Principal Investigator — Departement of obstetrics and gynecology, Linkopings University, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hjertberg L, Uustal E, Pihl S, Blomberg M. Maternal Body Mass Index and Anovaginal Distance in Active Phase of Term Labor. Biomed Res Int. 2018 Mar 7;2018:1532949. doi: 10.1155/2018/1532949. eCollection 2018. PMID 29707565